CLINICAL TRIAL: NCT02389842
Title: PIPA: a Phase Ib Study to Assess the Safety, Tolerability and Efficacy of the PI3K Inhibitors, Taselisib (GDC-0032) or Pictilisib (GDC-0941), in Combination with PAlbociclib, with the Subsequent Addition of Fulvestrant in PIK3CA-mutant Breast Cancers
Brief Title: PIPA: Combination of PI3 Kinase Inhibitors and PAlbociclib
Acronym: PIPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Roche Pharma AG (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4191; 2014-002658-37 (EudraCT Number)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2019-11

CONDITIONS: Advanced Solid Tumours; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palbociclib + Taselisib (Experimental): The starting dose of palbociclib in combination with taselisib will be 100mg OD of palbociclib and 2mg taselisib OD, administered orally 21-days-on and 7-days-off, as part of a 28 day cycle.
  Interventions: Drug: Palbociclib + Taselisib / Pictilisib
- Palbociclib + Pictilisib (Experimental): The starting dose of palbociclib in combination with pictilisib will be 100mg OD of palbociclib and 195 mg pictilisib OD, administered orally 21-days-on and 7-days-off, as part of a 28 day cycle.
  Interventions: Drug: Palbociclib + Taselisib / Pictilisib

INTERVENTIONS:
Drug: Palbociclib + Taselisib / Pictilisib

SUMMARY:
Part A: This is a phase Ib trial combining the CDK4/6 inhibitor palbociclib with the PI3K inhibitors taselisib, or pictilisib. There are two treatment arms during the dose escalation phase where patients will receive either taselisib OR pictilisib in combination with palbociclib. Palbociclib, taselisib and pictilisib can all be given orally once daily with food, in a 21-days-on and 7-days-off schedule. Once the MTD is reached, the combination with the optimum safety and PK/PD profile will be taken forward to the dose expansion phase (Part B).

Part B1: At the MTD dose expansion, fulvestrant will be administered in addition to palbociclib and taselisib or pictilisib orally once daily, in a 21-days-on and 7-days-off schedule in the ER+ve HER2-ve PIK3CA mutant breast cancer cohort. Fulvestrant will be given intramuscularly on Day 1, Day 15 in cycle one followed by Day 1 for all subsequent cycles.

Part B2: At the MTD dose expansion, patients with PIK3CA mutant advanced solid tumours will be treated with palbociclib and taselisib or pictilisib orally once daily, in a 21-days-on and 7-days-off schedule.

DETAILED DESCRIPTION:
This is a phase Ib trial of palbociclib in combination with either taselisib or pictilisib. The study will include a dose escalation phase (Part A), and an MTD dose expansion phase (Part B).

Part A: will investigate escalating doses of palbociclib with either pictilisib or taselisib administered orally, continuously for 21 days out of a 28 day cycle in patients with advanced solid tumours recruited simultaneously into two parallel arms (up to 24 patients in each arm with a maximum of 48 patients in Part A).

Once the MTD is determined the combination with the optimum safety and PK/PD profile as determined by the SRC will be taken forward to the dose expansion phase (Part B).

Part B: The MTD dose expansion phase will be conducted using the optimal combination from Part A in two parallel arms as follows:

B1: Patients (n=25) with PIK3CA mutant ER + HER2-ve advanced breast cancers will be treated with a triplet combination of palbociclib and either taselisib or pictilisib along with fulvestrant. Part B1 will require at least two of the first 15 patients to respond to progress to recruit the full 25 patients.

B2: Patients (n=20) with PIK3CA mutant advanced solid tumours including at least 8 patients with PIK3CA mutant ER negative and/or HER2 positive breast cancers will be treated with the doublet combination of palbociclib and either taselisib or pictilisib. Other cancers with relevant genetic aberrations (e.g. KRAS mutations) may be considered, depending on emerging preclinical and clinical data on these novel antitumour agents.

In total, it is expected that a minimum of 70 and up to a maximum of 93 patients will be enrolled into the trial, the final number will depend on the number of dose escalations required to reach DLT. If < 48 patients are enrolled in Part A, investigators will be permitted to enrol > 45 patients in Part B, providing the maximum number of patients remains ≤93 patients across the study.

The anticipated accrual rate during the dose escalation phase is estimated at 2 patients per month. Accrual in the expansion phase is estimated at 4 patients per month across 2 centres. It is expected that the trial will have a duration of recruitment of 12 to 24 months.

ELIGIBILITY:
Inclusion Criteria

1. Part A (dose escalation):

   Patients with histologically or cytologically confirmed malignant advanced solid tumours refractory to standard therapy or for which no suitable effective standard therapy exists, including, but not limited to patients with PIK3CA mutant cancers, or those with somatic mutations or other aberrations known to result in a hyperactivated PI3K-AKT pathway.

   Advanced breast cancer with the following features:
   * ER+ve breast cancer that has progressed on at least one line of prior endocrine therapy, or
   * PIK3CA mutant breast cancer progressed on at least one line of prior endocrine therapy or chemotherapy
   * breast cancer refractory to standard treatment

   Part B (dose expansion):

   Part B1 Patients with histologically or cytologically confirmed advanced ER+ve, HER2-ve breast cancer with a PIK3CA mutation confirmed by an accredited laboratory.

   Part B2
   * Patients with histologically or cytologically confirmed advanced solid tumours with mutations leading to a hyperactivated PI3K-AKT pathway, or other relevant genetic aberrations; OR
   * Patients with histologically or cytologically confirmed advanced ER-ve, HER2+ve breast cancer with a PIK3CA mutation confirmed by an accredited laboratory; OR
   * Patients with histologically or cytologically confirmed advanced triple negative breast cancer with a PIK3CA mutation confirmed by an accredited laboratory.

   Part B3 Patients with histologically or cytologically confirmed advanced ER+ve, HER2-ve breast cancer.

   NB. PIK3CA mutation may be assessed in archival tumour samples, fresh tumour samples, or in circulating free DNA extracted from plasma or serum and the result must be from an accredited laboratory. This is mandatory for breast cancer patients in Part B1 and B2 and the result must be available prior to the patient entering the main study.

   A mutation will be considered pathogenic if described to be recurrent somatic mutation in COSMIC (http://cancer.sanger.ac.uk/cancergenome/projects/cosmic/). Other cancers with relevant genetic aberrations (e.g. KRAS mutations) may be considered, depending on emerging preclinical and clinical data on these novel antitumour agents.
2. Prior cancer treatment as follows:

   * Patients with ER+ve and HER2-ve breast cancer in Parts B1 and B3 should have progressed on at least one prior hormone therapy and had a maximum of two prior lines of chemotherapy for advanced breast cancer;
   * Patients in the solid tumour AND triple negative breast cancer cohort of Part B2 must have progressed on at least one prior chemotherapy regimen for advanced cancer;
   * Patients with HER2+ve breast cancer in Part B2 should have progressed on at least two prior HER2 directed therapies for advanced breast cancer (or one prior therapy where no further HER2 directed therapy is available locally).
3. Part A: Measurable disease as assessed by RECIST 1.1 OR evaluable disease. Part B1: Measurable disease as assessed by RECIST 1.1 Part B2 and B3: Measurable disease as assessed by RECIST 1.1 OR evaluable disease
4. Life expectancy of at least 12 weeks
5. World Health Organisation (WHO) performance status of 0-1 with no significant deterioration over the previous 2 weeks (Appendix 1)
6. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.

Laboratory Test Value required Haemoglobin (Hb) ≥ 10.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 150 x 109/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with documented Gilberts' disease Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible

Creatinine - If creatinine > 1.5 times ULN then: Either:

Calculated creatinine clearance

Or:

Isotope clearance measurement

≤1.5 times ULN

* 50 mL/min (uncorrected value)
* 50mL/min (corrected) Coagulation INR <1.5, APTT <1.5x ULN

Exclusion criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous 4 weeks (6 weeks for nitrosoureas, Mitomycin-C) and 4 weeks for investigational medicinal products before treatment

   Exceptions to this are:
   * patients progressing on letrozole or fulvestrant;
   * hormonal therapy with luteinizing hormone-releasing hormone (LHRH) analogues for medical castration in patients with castrate resistant prostate cancer;
   * bisphosphonates or RANK ligand antagonists that are permitted for the management of bone metastases;
   * palliative radiotherapy if given for bony metastases, as long as these are not indicative of disease progression. Study drug must be stopped 3 days before radiotherapy and restarted within 28 days, as long as bone marrow function has returned to normal.
2. Patients with prior exposure to either a CDK4/6 inhibitor OR a PI3K/ATK/mTOR inhibitor are excluded from the study With the exception of allosteric mTOR inhibitors such as everolimus that is allowed. Prior exposure to fulvestrant or aromatase inhibitors is permitted.
3. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   * Diagnosis of diabetes mellitus types I or II (irrespective of management).
   * Glycosylated haemoglobin (HbA1C) ≥7.0% at screening
   * Fasting Plasma Glucose ≥ 6.9mmol/L at screening. Fasting is defined as no caloric intake for at least 8 hours.
4. On-going toxic manifestations of previous treatments ≥ grade 1. Exceptions to this are alopecia or certain other toxicities, which in the opinion of the Investigator should not exclude the patient.
5. History of malabsorption syndrome or other condition that would interfere with enteral absorption. For example active intestine inflammation (e.g., Crohn's disease or ulcerative colitis) requiring immunosuppressive therapy.
6. History of inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis)
7. Inability or unwillingness to swallow pills, or (for patients receiving fulvestrant) receive IM injections.
8. Known untreated or active central nervous system (CNS) metastases (progressing or requiring corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

   * Evaluable or measurable disease outside the CNS is present.
   * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the baseline disease assessment for at least 28 days.
   * Not requiring dexamethasone treatment.
9. Major surgery (excluding minor procedures, e.g. placement of vascular access) within 4 weeks of the first dose of study treatment.
10. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
11. Male patients with partners of childbearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.

    NB: Male patients who are potentially fertile should be made aware that palbociclib causes testicular degeneration in animal models and may wish to consider sperm preservation prior to beginning therapy.
12. At high medical risk because of severe or uncontrolled systemic disease, such as:

    uncontrolled hypertension, symptomatic congestive heart failure ≥ class 2 (refer to appendix 4 for grading), unstable angina pectoris, stroke or myocardial infarction within 6 months, serious cardiac arrhythmia requiring treatment, with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia or conduction abnormality that has been treated and for which the patient is no longer at risk for serious arrhythmia (e.g., Wolff-Parkinson-White syndrome treated with surgical ablation).
13. Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with hepatitis B virus, or hepatitis C virus.

    Active infection is defined as requiring treatment with antiviral therapy or presence of positive test results for Hepatitis B (Hepatitis B surface antigen [HBsAg] and/or total Hb core antibody [anti-HBc]) or Hepatitis C (Hepatitis C virus [HCV] antibody). Unless required by local regulations, patients are not required to have HIV, HCB, or HCV assessments at screening if these assessments have not been previously performed.

    Patients who are positive for anti-HBc are eligible only if testing is also positive for Hepatitis B surface antibody [HbsAb] and polymerase chain reaction (PCR) is negative for HBV DNA.

    Patients who are positive for HCV serology are eligible only if testing for HCV RNA is negative.
14. Immunocompromised status due to current known active infection with HIV or due to the use of immunosuppressive therapies for other conditions.
15. Need for current chronic corticosteroid therapy, specifically dexamethasone or ≥ 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids. Stable use (i.e., no change in dose within 1 month prior to Day 1 of Cycle 1) of inhaled corticosteroids is allowed.
16. Prior bone marrow transplant or extensive radiotherapy to greater than 25% of bone marrow within eight weeks.
17. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study. Participation in an observational trial would be acceptable.
18. Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 3 years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
19. Patients who require daily supplemental oxygen
20. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Recommended dose for Phase II | duration of study (24 months)
  To determine a dose at which no more than one patient out of up to six patients at the same dose level experience a highly probable or probable drug-related dose limiting toxicity.
Safety and Toxicity Profile (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0) | duration of study (24 months)
  To evaluate causality of each adverse event to palbociclib with taselisib and fulvestrant; palbociclib and taselisib; letrozole, palbociclib and taselisib against CTCAE criteria V4.0
Preliminary anti-tumour assessment of triplet combination (RECIST criteria version 1.1) in patients with PIK3CA mutant advanced ER+ve HER2-ve breast cancer. | duration of study (24 months)
  To evaluate disease response by RECIST criteria version 1.1, clinical benefit rate, best change in tumour size, progression free survival, and duration or response.

SECONDARY OUTCOMES:
Pharmaockinetics Profile (AUC0-24 and Cmax) | duration of study (24 months)
  To determine the plasma levels of the investigational drugs using validated assays: AUC0-24 and Cmax.

OTHER OUTCOMES:
Preliminary anti-tumour assessment (RECIST criteria version 1.1) of combinations. | duration of study (24 months)
  To evaluate disease response by RECIST criteria version 1.1, clinical benefit rate, best change in tumour size, progression free survival, and duration or response.
Mechanisms of Drug Resistance (deep sequence tumour and circulating tumour DNA) | duration of study (24 months)
  To deep sequence tumour and circulating tumour DNA at baseline, during treatment and on progression.
Pharmacodynamics of Pre- and Post-treatment tumour biopsies (biomarker changes) | duration of study (24 months)
  To determine biomarker changes, including: phospho (e.g. pRbser780) and total retinoblastoma protein (Rb), phospho (pSer473) and total AKT, phospho (pThr246) and total PRAS40, Ki67 and TUNEL.
Pharmacodynamics Profile using PRP (biomarker changes) | duration of study (24 months)
  To determine PD biomarker changes, such as: phospho and total AKT, GSK3b, pS70S6K and PRAS40 using the validated MSD electrochemiluminescent triplex platform.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Turner, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (2):
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Pascual J, Lim JSJ, Macpherson IR, Armstrong AC, Ring A, Okines AFC, Cutts RJ, Herrera-Abreu MT, Garcia-Murillas I, Pearson A, Hrebien S, Gevensleben H, Proszek PZ, Hubank M, Hills M, King J, Parmar M, Prout T, Finneran L, Malia J, Swales KE, Ruddle R, Raynaud FI, Turner A, Hall E, Yap TA, Lopez JS, Turner NC. Triplet Therapy with Palbociclib, Taselisib, and Fulvestrant in PIK3CA-Mutant Breast Cancer and Doublet Palbociclib and Taselisib in Pathway-Mutant Solid Cancers. Cancer Discov. 2021 Jan;11(1):92-107. doi: 10.1158/2159-8290.CD-20-0553. Epub 2020 Sep 21. PMID 32958578